CLINICAL TRIAL: NCT06960681
Title: Evaluation of the External Validity of the Knee SFA Score for the Detection of LCA Lesions in Emergency Departments
Brief Title: Evaluation of the External Validity of the Knee SFA Score
Acronym: SCORESFA
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0102/OB; IDRCB 2023-A02760-45 (Other: ANSM)
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-01

CONDITIONS: Reliability in the Detection of ACL Injuries in Emergency Departments
Keywords: ACL (anterior cruciate ligament)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: External validity of the SFA score — Testing the external validity of the SFA score for the detection of in adult emergency departments

SUMMARY:
A screening score for ACL (anterior cruciate ligament) injuries based on questioning has been developed by the Société Francophone d'Arthroscopie to provide better guidance for post-trauma patients. The score differentiates between 3 groups of patients: mild trauma (score 1 to 4), intermediate trauma (score 5 to 7) and severe trauma (score 8 to 12).

The main hypothesis of this study is that it is a reliable score for detecting ACL injuries in emergency departments.

DETAILED DESCRIPTION:
Injury to the anterior cruciate ligament is a serious and not uncommon event, which can affect the functional future of the knee. The result is instability, leading to meniscal and osteo-cartilaginous damage in the medium and long term. Early diagnosis would limit the occurrence of these complications.

The average annual incidence of ACL rupture in the French population is estimated at around population can be estimated at around 0.03%, or approximately 20,000 cases per year. Diagnosis is currently based on clinical examination and dynamic ligament testing. However, these may be difficult to perform in the immediate post-trauma period, leading to a delay in diagnosis. Magnetic resonance imaging (MRI) is a good diagnostic tool, with a sensitivity of 83-95% and a specificity of 95-100%. However, access to MRI is still limited in emergencies, with an average appointment time (all indications combined) of 32.3 days. It is therefore to better target the indications for this examination.

The Société Francophone d'Arthroscopie has developed a screening score for ACL lesions, based on questioning, to help guide post-trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to adult emergency departments with knee trauma less than 9 days old;
* All patients aged between 18 and 55;
* All patients without an X-ray fracture (with the exception of indirect signs of injury to the central pivot: Segond's fracture and avulsion of the tibial spines);
* All patients affiliated to or benefiting from a social security scheme;
* All patients who have given their and who have received a study information sheet.

Exclusion Criteria:

* Trauma requiring immediate surgical treatment (fracture, dislocation);
* Previous osteoarticular trauma to the knee;
* Pregnant women;
* Impossible to carry out an MRI (contraindication, refusal, claustrophobia);
* Impossible to provide follow-up in the same centre;
* Protected patients: adults under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient with a rupture of the anterior cruciate ligament (ACL) diagnosed during a follow-up visit to the emergency department (diagnosed on clinical examination and/or MRI) and with a score ≥ 8.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
External validity of the SFA score | At enrollment visit, Month 1
  Testing the external validity of the SFA score for the detection of in adult emergency departments

SECONDARY OUTCOMES:
Sensitivity of the different score items (EVA > 6) | At enrollment visit, Month 1
  Analyse the sensitivity of the EVA score for screening for ACL injuries (EVA > 6)
Sensitivity of the different score items (functional impotence > 1) | At enrollment visit, Month 1
  Analyse the sensitivity of the functional impotence score for screening for ACL injuries (functional impotence > 1)
Sensitivity of the different score items (Cracking ≥ 1) | At enrollment visit, Month 1
  Analyse the sensitivity of the Cracking score for screening for ACL injuries (Cracking ≥ 1)
Sensitivity of the different score items (Instability ≥ 1) | At enrollment visit, Month 1
  Analyse the sensitivity of the Instability score for screening for ACL injuries (Instability ≥ 1)
Sensitivity of the different score items (Presence of an effusion) | At enrollment visit, Month 1
  Analyse the sensitivity of the effusion score for screening for ACL injuries (Presence of an effusion)
Specificity of the different score items (EVA > 6) | At enrollment visit, Month 1
  Analyse the Specificity of the EVA score for screening for ACL injuries (EVA > 6)
Specificity of the different score items (functional impotence > 1) | At enrollment visit, Month 1
  Analyse the Specificity of the functional impotence score for screening for ACL injuries (functional impotence > 1)
Specificity of the different score items (Cracking ≥ 1) | At enrollment visit, Month 1
  Analyse the Specificity of the Cracking score for screening for ACL injuries (Cracking ≥ 1)
Specificity of the different score items (Instability ≥ 1) | At enrollment visit, Month 1
  Analyse the Specificity of the Instability score for screening for ACL injuries (Instability ≥ 1)
Specificity of the different score items (Presence of an effusion) | At enrollment visit, Month 1
  Analyse the Specificity of the effusion score for screening for ACL injuries (Presence of an effusion)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan JC CURADO, Doctor, Study Director — Service de Chirurgie Orthopédique et Traumatologie, UH Rouen
Locations (3):
- France (3):
  - Groupe Hospitalier du Havre J. Monod, Montivilliers
  - University Rouen Hospital, Rouen
  - University Hospital of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.